CLINICAL TRIAL: NCT02116738
Title: Interventional Study of the Relatively New Surgical Techniques on the Treatment of Pilonidal Sinus Disease
Brief Title: Modified Limberg Procedure Versus Lateral Advancement Flap With Burrow's Triangle Procedure in the Treatment of Pilonidal Sinus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Mevki Military Hospital (Other)
Responsible Party: Principal Investigator, MD. Mehmet SAYDAM (General Surgeon), MD. MEHMET SAYDAM (GENERAL SURGEON), Ankara Mevki Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMMA-LEC-001642
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Sacrococcygeal Pilonidal Disease
Keywords: flap; pilonidal sinus; vas; recurrence
MeSH Terms: conditions — Pilonidal Sinus; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flap Transposition Technique (Experimental): Flap Transposition Technique
  Interventions: Procedure: Flap Transposition Procedures

INTERVENTIONS:
Procedure: Flap Transposition Procedures — Modified Limberg Flap Transposition Procedure and Lateral Advancement Flap Transposition with Burrow's Triangle Procedure in The treatment of Pilonidal Sinus Diseases

SUMMARY:
The investigators want to share our study that is the "Comparison of Modified Limberg Flap Transposition and Lateral Advancement Flap Transposition with Burrow's Triangle in the Surgical Treatment of Sacrococcygeal Pilonidal Sinus.

DETAILED DESCRIPTION:
Pilonidal Sinus Disease (PSD) is a common and chronic entity of the young adults. So far, many options regarding the surgical treatment of the disease has been described, the consensus about treatment stills remains unsatisfactory, as all the surgical methods have encountered with different rate of recurrences. Our aim in this study is to compare the widely used technique in pilonidal sinus surgical treatment Modified Limberg Flap Transposition and relatively less used technique Lateral Advancement Flap Transposition with Burrow's Triangle, in the terms of VAS scores, recurrence, postoperative complications, surgical site infections in the first 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pilonidal Sinus Disease
* Must be able to suitable for the surgery

Exclusion Criteria:

* Patients with Recurrent Pilonidal Sinus disease
* Patient whom is not suitable for surgery

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a 95% Decrease in Pain Visual Analogue Scale (VAS) | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Mevki Military Hospital : General Surgery Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Yuksel BC, Berkem H, Ozel H, Hengirmen S. A new surgical method of pilonidal sinus treatment: a bilaterally paralel elliptic fascio-cutaneous advancement flap technique. Bratisl Lek Listy. 2012;113(12):728-31. doi: 10.4149/bll_2012_165. PMID 23173633
- See also: Turkish Surgical Association — http://turkcer.org.tr